CLINICAL TRIAL: NCT01705262
Title: Comparing Oral Preparation With Macrogol (Moviprep) and Natriumdihydrogenphosphatdihydrat (Phosphoral)
Status: Terminated | Type: Observational
Why Stopped: Phophoral was no longer used as a preparation before coloscopies at OUH
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anne Reiss Axelsen, MD, Odense University Hospital
Other Study IDs: AAX-001
Record Dates: First submitted 2012-01-27; First posted 2012-10-12 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Colonoscopy
Keywords: compliance; Bowel preparations; Moviprep; Phosphoral
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- u-65 M: Male patients under 65
- u-65 K: Female patients under 65 years old
- o-65 -K: Female patients over 65 years
- O-65 M: Male patients over 65 years

SUMMARY:
The purpose of this study is to determine whether Moviprep or Phosphoral is the best method of bowel preparation before colonoscopy - seen by the patients and by the endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnostic colonoscopy,
* colonoscopy as a follow-up,
* intended therapeutic colonoscopy.

Exclusion Criteria:

* patients younger than 18 years
* pregnancy
* known bowl obstructions
* known inflammatory colon disease
* known kidney disease
* phenylketonuri
* glucose-6-phospat deficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to colonoscopy by the house doctors
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Surgery department, Odense, Odense, Denmark